CLINICAL TRIAL: NCT07352657
Title: Remote Alert Pathway To Optimize CaRe of Cardiac Implantable Electrical Devices: The RAPTOR-CIED Study (Main Phase)
Acronym: RAPTOR - MAIN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Daniel B. Kramer, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025P001064
Record Dates: First submitted 2026-01-12; First posted 2026-01-20 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Pacemaker; Implantable Defibrillator

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Guideline-based Care (Active Comparator): Remote monitoring programming scheduled for alert transmissions, patient-initiated transmissions, and routine transmissions (scheduled to occur every 90 days from the date of enrollment in the study); in-office interrogations on at least an annual basis
  Interventions: Other: Guideline-based Care
- Alert-based care (Active Comparator): Alert-based care is an alternative strategy for longitudinal management of patients with wireless pacemakers and implantable defibrillators
  Interventions: Other: Alert-based care

INTERVENTIONS:
Other: Alert-based care — Alert-based care is an alternative strategy for longitudinal management of patients with wireless pacemakers and implantable defibrillators
  Arms: Alert-based care
Other: Guideline-based Care — Remote monitoring programming scheduled for alert transmissions, patient-initiated transmissions, and routine transmissions (scheduled to occur every 90 days from the date of enrollment in the study); in-office interrogations on at least an annual basis
  Arms: Guideline-based Care

SUMMARY:
he Remote Alert Pathway to Optimize Care of Cardiac Implantable Electrical Devices (RAPTOR-CIED) Study is a pragmatic, multi-center, randomized trial with 1:1 patient-level randomization comparing the safety and effectiveness of alert-driven care versus guideline-based care for patients with wireless cardiac implantable electrical devices (CIEDs).

The study will be conducted in 2 phases: a Feasibility Phase and a Main Phase. This registration outlines the goals and design features of the Main Phase of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged > 18 years
2. Clinically stable by investigator assessment
3. Has a newly implanted or existing wireless CIED: single, dual-chamber, biventricular, subcutaneous/extravascular, and leadless systems are all eligible, including pacemakers or implantable cardioverter-defibrillators (ICDs)
4. CIED is from one of the 4 major CIED manufacturers in the US market (99% of implants in the US): Medtronic, Boston Scientific, Abbott, Biotronik
5. Currently enrolled in remote monitoring as part of standard of care
6. Primary clinical electrophysiology follow-up at the enrolling center
7. Understands spoken and written English, Spanish, or Portuguese
8. Has sufficient cognitive function to answer standardized questions about study rationale and procedures.

Exclusion Criteria:

1. Presence of insertable cardiac monitor, either in isolation or in combination with any other CIED
2. Listed for cardiac transplantation prior to enrollment (N.B. if a patient becomes listed for transplantation during the study, they may continue study participation)
3. Participation in another study related to novel CIED technology or remote monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-01-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events | 2 years
  Incidence of MACE (i.e., death, stroke or systemic embolism, and unplanned cardiac device procedure)
Effectiveness | 2 Years
  Proportion of total device related encounters that are actionable (e.g., changes in programming or treatment)

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided